CLINICAL TRIAL: NCT03454061
Title: The Development of Motor Skills by a Physical Education Programme in Preschool Children: a Preschool-based Controlled Trial
Brief Title: Effects of a Physical Education Programme in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Giuseppe Battaglia, PhD, University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH Project
Record Dates: First submitted 2018-02-07; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Motor Activity; Child Development
Keywords: sport; physical activity; education; fundamental motor skills; childhood; exercise; health; training; intervention; gross motor development
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Physical activity intervention
  Interventions: Other: physical activity
- Control (No Intervention): Keep usual activities in kindergarten

INTERVENTIONS:
Other: physical activity — Physical education program (PEP) of 16-week length
  Arms: Intervention

SUMMARY:
Unlike other European countries, Italian kindergartens do not include the physical education teacher in the school organic personnel. This is frequently associated with the lack of opportunities to perform physical education by preschool children. The aim of this study was to analyse the effects of a specific 16-week-long physical education programme (PEP) of 16-week length on the development of locomotor and object control skills in preschool children.

DETAILED DESCRIPTION:
We conducted a school-based non-randomised controlled trial to evaluate the effect of a specific 16-week-long physical education program (PEP) on the quotient of gross motor development (QGMD) in preschool children. This study involved 119 children who were clustered in a control group (CG, n= 29, age: 52.1±8.65 months; height: 1.1±0.07 m, body weight: 19.2±5.55 Kg, BMI: 16.9±3.16) and an intervention group (IG, n= 90, age: 57.4±9.42 months; height: 1.1±0.06 m, body weight: 19.3±3.65 Kg, BMI: 16±1.75). Participants were assessed for locomotor ability and object control skills using the Italian version of gross motor development test, before and after the experimental period.

ELIGIBILITY:
Inclusion Criteria

* preschool children

Exclusion Criteria:

* Age < 40 months
* Age > 67 months

Ages: 40 Months to 67 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Quotient of gross motor development change | Change from Baseline at 16 weeks
  Quotient of gross motor development

SECONDARY OUTCOMES:
BMI | Change from Baseline at 16 weeks
  Body mass index
Weight | Change from Baseline at 16 weeks
  Weight
Height | Change from Baseline at 16 weeks
  Height
Object control skills change | Change from Baseline at 16 weeks
  Object control
Locomotion skills change | Change from Baseline at 16 weeks
  locomotion

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Bellafiore, Study Director — University of Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tabacchi G, Battaglia G, Alesi M, Paoli A, Palma A, Bellafiore M. Food literacy predictors and associations with physical and emergent literacy in pre-schoolers: results from the Training-to-Health Project. Public Health Nutr. 2020 Feb;23(2):356-365. doi: 10.1017/S1368980019002404. Epub 2019 Sep 2. PMID 31474231